CLINICAL TRIAL: NCT05817929
Title: Angiopoietin Dysregulation to Predict Adverse Outcomes in Cardiac Surgery: the Prospective
Brief Title: Angiopoietin and Adverse Outcomes in Cardiac Surgery
Acronym: ANGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0015
Record Dates: First submitted 2023-03-23; First posted 2023-04-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery; Acute Kidney Injury
Keywords: angiopoietin; endothelial injury; MACCE
MeSH Terms: conditions — Acute Kidney Injury | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cardiac surgery (Experimental)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — 5 ml blood sample will be withdrawn at the surgery start and at the surgery end

SUMMARY:
Cardiac surgery and cardiopulmonary bypass can lead to systemic organ failure trough excess inflammation and endothelial injury. The angiopoietin family represented by angiopoietin 1 and 2 can reflect endothelial injury by a decrease in angiopoietin 1 and an increase in angiopoietin 2. The investigators hypothesized that angiopoietin dysregulation could reflect organ failure related to cardiac surgery.

The purpose of this project is to assess the association between angiopoietin dysregulation and adverse outcomes on cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patient scheduled for cardiac surgery under cardiopulmonary bypass

Exclusion Criteria:

* patient less than 18 years old,
* redo surgery,
* urgent surgery,
* endocarditis,
* aortic root repair surgery
* aortic dissection
* heart beating surgery,
* heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Correlation between abnormal angiopoietin 1 concentration (ng/ml) and number of major cardiovascular event | 28 days
  major cardiovascular event are myocardial infraction, stroke, acute kidney injury, cardiovascular death
correlation between occurence of abnormal angiopoietin 2 concentration (ng/ml) and occurence of major cardiovascular event | 28 days
  major cardiovascular event are myocardial infraction, stroke, acute kidney injury, cardiovascular death

SECONDARY OUTCOMES:
Correlation between abnormal angiopoietin 1 concentration (ng/ml) and number of postoperative pulmonary complications | 28 days
Correlation between abnormal angiopoietin 2 concentration (ng/ml) and number of postoperative pulmonary complications | 28 days
Correlation between abnormal angiopoietin 1 concentration (ng/ml) and mortality at 3 months | 3 months
Correlation between abnormal angiopoietin 2 concentration (ng/ml) and mortality at 3 months | 3 months
Correlation between abnormal angiopoietin 1 concentration (ng/ml) and mortality at 6 months | 6 months
Correlation between occurence of abnormal angiopoietin 2 concentration (ng/ml) and mortality at 6 months | 6 months
Correlation between abnormal angiopoietin 1 concentration (ng/ml) and mortality rate at 12 months | 12 months
Correlation between abnormal angiopoietin 2 concentration (ng/ml) and mortality rate at 12 months | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No